CLINICAL TRIAL: NCT05441696
Title: Pilot Study for the Evaluation of EzCVP in Heart Failure Patients
Brief Title: Study for the Evaluation of a Non-invasive Hemodynamic Measurement in Heart Failure Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Nihon Kohden (Industry)
Responsible Party: Sponsor
Other Study IDs: 70Ag_Ogino-00026
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-03

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Adult CHF subjects with initial high CVP: Adult subjects with congestive heart failure diagnosis who have an indicated high non-invasive estimated central venous pressure on first measurement after clinical unit admission.
  Interventions: Device: ezCVP measurement
- Adult CHF subjects with initial low CVP: Adult subjects with congestive heart failure diagnosis who have an indicated low non-invasive estimated central venous pressure on first measurement after clinical unit admission.
  Interventions: Device: ezCVP measurement

INTERVENTIONS:
Device: ezCVP measurement — * Measuring device: non-FDA-cleared patient monitor (740E, Zoe Medical, MA, US), which has software to measure ezCVP.
  * Sensor: an FDA-cleared pulse oximeter sensor for adults (K012891: DS-100A, Nellcor, CA, US).
  * Cuff: an FDA-cleared NIBP cuff for adults (K080342: YP-713T, YP-714T or TP-715T, Nihon Kohden Corporation, Tokyo, Japan).

SUMMARY:
Track changes in non-invasive central venous pressure across hospital stay and relationship with readmission

DETAILED DESCRIPTION:
Determining the degree of congestion is important in deciding appropriate timing for discharging hospitalized heart failure patients. Central venous pressure (CVP) reflects the returning blood volume to the heart and can guide therapy to relieve congestion. However, the conventional method used to measure CVP has notable limitations as it is an invasive procedure that requires placement of a central venous catheter.

Traditional, non-invasive methods of estimating CVP, such as physical examination and echocardiogram, are less accurate and more resource intensive. To overcome this challenge, new technology to assess CVP non-invasively using an oscillometric method has been developed. This new technology involves measurement of the enclosed zone central venous pressure (ezCVP), which, in a preclinical study, has been shown to correlate with invasive data.

Additionally, a previous correlation study demonstrated that the ezCVP value can be mathematically adjusted to estimate invasive CVP. The resulting value has been termed CVPNI (CVP Non-Invasive). Most recently, a limited pilot study of patients hospitalized with acute, decompensated heart failure demonstrated the feasibility of device use in this population and the expected and incremental fall in CVPNI with medical treatment over the course of hospitalization.

Moving forward, and in order to further improve the care of patients hospitalized with heart failure, an expanded pilot study of ezCVP technology is needed to prove that changes in CVPNI track with these patients' condition during admission and can be useful in their clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Arm circumference of 23 cm to 55 cm
* Subject admitted to the hospital with acute exacerbation of heart failure, with either reduced or preserved ejection fraction
* Subject is at risk for readmission (NYHA Functional Classification 2-3)
* Subject is able to understand the risks and potential benefits of participating in the study and is willing to provide written, informed consent
* ezCVP indicator is high (CVPNI is over 9 mmHg) at admission
* Subject is willing and able to comply with protocol procedures
* Subject tested negative for COVID test after admission to the hospital

Exclusion Criteria:

* Finger and upper arm anatomical anomaly or disease that may interfere with attaching a pulse oximeter sensor and/or blood pressure cuff
* Pregnant (self-reported)
* Upper extremity DVT (currently being treated)
* Severe skin disease involving the upper arm(s)
* Study investigator may exclude patients based on clinical judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted due to heart failure exacerbation
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Evaluate the difference between non-invasive CVP measurement at admission and at discharge | 7 days
  Compare CVPNI at time of admission and discharge in clinical unit CVPNI (CVP subscript NI) is a numeric value equivalence of central venous pressure non-invasive measured in mmHg.
Evaluate the difference between non-invasive CVP measurement in right and left arms | 7 days
  Compare CVPNI (mmHg) for measurements on left and right arm for same subject

SECONDARY OUTCOMES:
Evaluate the relationship between CVPNI at discharge and readmission rate | 100 days
  Compare CVPNI (mmHg) at time of discharge for high ezCVP subjects to subsequent readmission occurrence within 90-100 days post hospital discharge
Evaluate the relationship between CVPNI to clinical parameter weight during hospitalization | 7 days
  Compare CVPNI changes (∆ mmHg) for high ezCVP subjects during hospitalization to change in measured weight (∆ g)
Compare changes in CVPNI to changes in KCCQ quality scores | 21 days
  For each of the 3 Kansas City Cardiomyopathy Questionnaire (KCCQ) totals (integer number with no unit of measure): 1. Overall summary score; 2. clinical summary score; 3. symptom stability score: calculate: ∆KCCQ = KCCQ@14 days - KCCQ@admission. Count number of subjects in each group: ABSOLUTE(∆KCCQ) < 6 (no significant change); ∆KCCQ >= 6 (significant change improvement); ∆KCCQ <= -6 (significant change worsening).
  Compare to ∆CVPNI (unit = mmHg) = CVPNI-mean@admission - CVPNI-mean@discharge. Count number of subjects in each group: ∆CVPNI <= 0 (no improvement or worsening); ∆CVPNI > 0 & < 5 (improvement); ∆CVPNI > 5 (large improvement).
Evaluate the relationship between CVPNI and readmission rate for low and high ezCVP subjects | 100 days
  Compare CVPNI at time of discharge for high ezCVP subjects versus low ezCVP subjects to subsequent readmission occurrence within 90-100 days post hospital discharge. Readmission is a binary value (true or false).

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Kawana, MD, Principal Investigator — Stanford University; Patricia Nguyen, MD, Principal Investigator — Veterans Affairs Hospital Palo Alto
Locations (2):
- United States (2):
  - Veterans Affairs Hospital, Palo Alto, California
  - Stanford Medical Center, Stanford, California

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Aggregate results will be published by the investigators in academic journals.